CLINICAL TRIAL: NCT06642233
Title: Relationships Among Cervical Functional Test in Patients With Unspecific Neck Pain: a Descriptive and Correlation Study
Brief Title: Mobility of the Cervical Spine in Patients With Unspecific Neck Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Katarzyna Wojnicz, Principal Investigator, Wroclaw University of Health and Sport Sciences
Other Study IDs: KWojniczWUHSS
Record Dates: First submitted 2024-06-23; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Manual Therapy; Cervical Spine; Neck Pain
Keywords: manual therapy; cervical spine; neck pain; unspecific neck pain; body composition; functional neck tests; craniovertebral angle; CROM
MeSH Terms: conditions — Neck Pain | interventions — Pain Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women and men aged 18-75: People with a medical diagnosis of unspecific pain in the cervical spine - acute and chronic pain, regardless of when it began.
  Interventions: Diagnostic Test: Socio-demographic survey; Diagnostic Test: Visual Analogue Scale; Diagnostic Test: The World Health Organization Quality-of-Life Scale-BREF questionnaire; Diagnostic Test: The International Physical Activity Questionnaire; Diagnostic Test: The Neck Disability Index questionnaire; Device: Body composition analysis using TANITA device; Diagnostic Test: Cervical spine AROM (Active range of motion); Diagnostic Test: Sagittal plane UCS AROM (Upper cervical spine active range of motion); Diagnostic Test: Flexion-Rotation Test; Diagnostic Test: Sidebending-Rotation Test; Diagnostic Test: Axial rotation test C0-C2; Diagnostic Test: Tilting test C0-C1 and C2-C3; Diagnostic Test: Craniocervical flexion test; Diagnostic Test: Craniovertebral angle

INTERVENTIONS:
Diagnostic Test: Socio-demographic survey — Socio-demographic survey includes: age, sex, time of symptoms, work activity, hours of work activity, work position, activities with loads, physical activity, household chores, missing teeth, dental splints, dentures, smoking, alcohol consumption, whether they can reproduce their symptoms, hours during which they perform focal distance tasks, whether they have visual problems, whether they take painkillers or anti-inflammatory drugs, presence of headaches and their frequency), whether you can reproduce your symptoms, hours during which you perform tasks at focal distance, whether you have visual problems, whether you take analgesics or anti-inflammatory drugs, presence and frequency of headaches.
Diagnostic Test: Visual Analogue Scale — VAS scale - The subject must indicate with a horizontal line their perception of pain on a scale (not numbered) of 100 millimetres, with 0 being the absence of pain and 100 the worst pain imaginable. The patient will complete the VAS scale, responding to the average, maximum and minimum pain experienced throughout its duration.
Diagnostic Test: The World Health Organization Quality-of-Life Scale-BREF questionnaire — The WHOQOL-BREF questionnaire is used to assess domains quality of life: physical, mental, social functioning and functioning in the environment. Responses are on a 5-point scale (score range 1-5). In each field you can get maximum 20 points. The results of individual areas are positive (the higher the number of points, the higher the quality of life).
Diagnostic Test: The International Physical Activity Questionnaire — The International Physical Activity Questionnaire (IPAQ) is a self-reported questionnaire for assessing physical activity and sedentary behavior for adults aged 15-69 years, across a range of socio-economic settings.
Diagnostic Test: The Neck Disability Index questionnaire — The NDI evaluates the effect of neck pain on activities of daily living and social relationships. It consists of 10 items with 6 response options that are scored from 0 to 5 points each for a total possible score of 50. The classification of disability is based on the total score obtained, with higher number indicating greater disability.
Device: Body composition analysis using TANITA device — TANITA device - body composition analyzer, the proportion of muscle mass and fat in the upper limbs
  * Body height will be determined using a SECA 217 stadimeter.
  * General and segmental body composition using the eight-electrode body composition analyzer by TANITA.
Diagnostic Test: Cervical spine AROM (Active range of motion) — Measurement of cervical spine AROM can be performed using the CROM system (Performance Attainment Associates, Roseville, MN, USA). Flexion, extension, side bending to the right and left, and rotation to the right and left of the cervical spine are examined.
  The CROM measuring equipment consists of a helmet-shaped structure with the shape of glasses. These glasses adjust to the nasal septum thanks to the velcro on the back to fit them on the head. Three inclinometers for measuring on 3 cardinal planes were placed in the plastic construction.
Diagnostic Test: Sagittal plane UCS AROM (Upper cervical spine active range of motion) — Measurement of sagittal plane UCS AROM can be performed using the CROM system. Flexion and extension of the upper cervical spine are examined.
Diagnostic Test: Flexion-Rotation Test — The flexion-rotation test can be performed using the CROM system. Rotation of the upper cervical spine is tested while the cervical spine is flexed.
Diagnostic Test: Sidebending-Rotation Test — The sidebending-rotation test can be performed using the CROM system. Rotation of the upper cervical spine is tested while the cervical spine is in a lateral tilt.
Diagnostic Test: Axial rotation test C0-C2 — The Axial rotation test C0-C2 can be performed using the CROM system. Rotation of the C0-C2 is examined.
Diagnostic Test: Tilting test C0-C1 and C2-C3 — The Tilting test C0-C1 and C2-C3 can be performed using a goniometer. Lateral tilt of the C0-C1 and C2-C3 are examined.
Diagnostic Test: Craniocervical flexion test — The test measures the level of activation of the deep neck flexors using a pressure biofeedback device, an air-filled manual pressure cuff (Stabilizer TM, Chattanooga Group, INC., USA).
Diagnostic Test: Craniovertebral angle — The test measure the craniovertebral angle using a telephone placed on a tripod and a computer program. The CVA measurement is defined as the angle a horizontal line passing the neural spine of C7 in relation to the line connecting the tragus and the neural spine of C7.

SUMMARY:
The goal of this clinical trials is to describe and correlate the posture, function and disability of the cervical spine in patients with unspecific neck pain. The research hypothesis is: In patients with unspecific neck pain, there is a significant correlation between posture, function and disability of the cervical spine. Participants will take part in functional tests and complete surveys and questionnaires.

DETAILED DESCRIPTION:
The increasing number of people working for a long time in one body position or performing physical work causes an increasing incidence of unspecific neck pain. This translates into an increased need for examination and rehabilitation of these patients. The gold standard for evaluating and treating these patients has yet to be established and current methods are not complete.

The complementary objectives of the researches will be to describe the craniovertebral angle, the range of motion of the cervical and upper cervical spine, deep flexor activation, disability, functional variables in the unspecific neck pain and the correlation of posture, function and cervical spine disability variables in the unspecific neck pain.

The study participants will be women and men aged 18 to 75 suffering from unspecific neck pain.

People who agree to participate in the study will receive information about the research project and its goals. Any interested person will have the opportunity to discuss any aspect of the research with the project leader. All participants are also reminded that their anonymity is guaranteed, that they can withdraw from the project at any time without giving any explanation and that the data obtained are for only research purposes. There will be no prior information about the division of participants into groups. Individuals who ultimately agree to participate in the study must sign an informed written consent.

All measurements will be performed in one room, where constant environmental conditions will be maintained during the procedure, which will increase the reliability, accuracy and validity of the research. The doctoral student - researcher will be responsible for contacting and setting the dates and times of the meeting with patients, as well as for the entire administrative procedure, such as: information documents, explanations, obtaining informed written consent to participate in the project. The assessment procedure and measurements will be carried out by the doctoral student. Participants will be informed that they may not share information about the measurement results and the intervention received with any of the other project participants in order to maintain their blinding.

The first condition for joining the study will be meeting the inclusion and exclusion criteria. Once the sample is selected, an initial assessment will be performed by collecting data on the patients history.

Project participants will take part in one study. During the study, the participant will complete the given questionnaires, the body composition analysis and then manual tests will be performed. Cervical spine safety tests will be performed prior to manual testing. The approximate duration of the assessment session will be 90 minutes.

The patient will be informed that the procedure must be painless at all times and only a feeling of tightness or stretching is acceptable (below 3 out of 10 on the VAS scale). The outline of the design study protocol is as follows:

1. Socio-demographic survey
2. VAS scale
3. The WHOQOL-BREF questionnaire
4. The IPAQ questionnaire
5. The Neck Disability Index questionnaire (NDI)
6. Body composition analysis using TANITA device
7. Cervical spine AROM
8. Sagittal plane UCS AROM
9. Flexion-Rotation Test
10. Sidebending-Rotation Test
11. Axial rotation test C0-C2
12. Tilting test C0-C1 and C2-C3
13. Craniocervical flexion test
14. Craniovertebral angle

ELIGIBILITY:
Inclusion Criteria:

* age 18-75 years
* medical diagnosis of non-specific pain in the cervical spine (M54.2 - neck pain) - acute and chronic pain, regardless of when it began
* negative result of cervical spine safety tests
* obtaining written consent to conduct research

Exclusion Criteria:

* pregnancy
* pacemaker
* active cancer
* no consent to conduct research
* difficulty communicating
* the presence of a metal plate in the head and metal screws in the body
* positive cervical spine safety test
* condition after operations in the area of the cervical spine
* condition after fractures in the cervical spine
* vascular abnormalities and pathologies resulting in symptoms of vertebrobasilar insufficiency (carotid artery occlusion or dissection, vertebral artery insufficiency, emboli)
* contraindications to manual therapy or exercise
* has participated in a cervical spine exercise or manual therapy program in the last three months
* present clear signs of having suffered a significant whiplash injury
* inability to maintain a supine position
* no possibility to perform a flexion-rotation test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients applying for individual therapy at the private manual medicine rehabilitation center (Łubinowa street 12/4, 52-210 Wrocław - Poland) and meeting the conditions for inclusion in the study group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical Range of Motion | Baseline
  The CROM (Performance Attainment Associates, Roseville, MN, USA) is a device used to measure degrees of range of motion (ROM) in the cervical spine. The CROM measuring equipment consists of a helmet-shaped structure with the shape of glasses. These glasses adjust to the nasal septum thanks to the velcro on the back to fit them on the head. Three inclinometers for measuring on 3 cardinal planes were placed in the plastic construction. The range of flexion, extension, lateral bending, and rotation will be measured in degrees.

SECONDARY OUTCOMES:
Pain intensity | Baseline
  The Visual Analog Scale (VAS) consists of a visual graduated scale from 0 to 10 cm, where 0 represents the absence of pain and 10 represents very intense pain, used to measure the pain experienced by the patient. The participant will complete the VAS scale, responding to the average, maximum and minimum pain experienced throughout its duration.
Quality of Life level | Baseline
  To assess the quality of life of the participants, the WHOQOL-BREF will be utilized, an abbreviated instrument developed by the World Health Organization. This questionnaire will consist of 26 items distributed across four main domains: Physical, Psychological, Social Relationships, and Environment. Each item will be rated on a 5-point Likert scale, ranging from 1 ("not at all") to 5 ("extremely"). The scores for each domain will be calculated from the averages of the corresponding item responses, multiplied by 4 to transform the results into a scale of 0 to 100. Higher scores will indicate a better perception of quality of life in the specific domain.
Degree of Functional Disability | Baseline
  The Neck Disability Index (NDI) questionnaire, which assesses the degree of functional disability of the cervical region, is a self-administered questionnaire consisting of 10 sessions with 6 responses, reflecting 6 stages of functional disability, with scores ranging from 0 to 5, where 0 represents the lowest and 5 represents the highest level of disability.
Physical activity level | Baseline
  Measured using the short version of the International Physical Activity Questionnaire (IPAQ). Questionnaire contains 7 questions about all types of physical activity related to everyday life, work and leisure. Results are reported in categories depending on the variable 'MET minutes a week'. MET minutes represent the amount of energy expended carrying out physical activity. High physical activity (one hour of more of physical activity per day), moderate physical activity (half an hour of physical activity per day) or low physical activity (not meeting any of the criteria for either moderate or high levels of physical activity).
Craniovertebral angle | Baseline
  The CVA measurement is defined as the angle a horizontal line passing the neural spine of C7 in relation to the line connecting the tragus and the neural spine of C7. Two markers are placed on the ground, 1.5 m apart, in which there is a camera or smartphone and the subject. Reference markers are placed on the C7 spinous process and the ear swallow of the examined person, which are identified by palpation. The subject is placed on a mark on the floor, barefoot and standing, facing the evaluator. The researcher then takes the photo. To measure the craniovertebral angle, a horizontal line is drawn starting from the spinous process of the seventh cervical vertebra using the angular dimension of the computer program. Then, an oblique line is drawn through the tragus of the ear to the spinous process of the seventh cervical vertebra. The craniovertebral angle is measured and will form where these 2 lines meet (spinous process of the 7th cervical vertebra).
Activation of the deep flexor muscles | Baseline
  The Stabilizer Pressure Biofeedback Unit (Chattanooga, TN, USA) is used for measurement. Activation and resistance of the deep cervical flexors are assessed in five progressive pressure increases from 2 mmHg to a maximum of 30 mmHg. When the patient reaches a level three times, they move on to the next level.
Body composition analysis | Baseline
  Body mass (Body composition analyzer BC 418 MA by Tanita), body height (height gauge SECA 217), based on them, determination of the BMI index and BMI percentile using percentile grids developed based on the OLAF program. Analysis of general and segmental parameters:
  * FatP - body fat mass in %,
  * FatM - body fat mass in kg,
  * FFM - body fat-free mass,
  * TBW - body water quantity in kg and %.
  * FFF index - based on the values of body fat and fat-free tissue, the general and segmental fat-free index is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Wojnicz, Master, Principal Investigator — Wroclaw University of Health and Sport Sciences
Locations (1):
- Wroclaw University of Health and Sport Sciences, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zarate-Tejero CA, Rodriguez-Rubio PR, Brandt L, Krauss J, Hernandez-Secorun M, Lucha-Lopez O, Hidalgo-Garcia C. Association between Age, Sex and Cervical Spine Sagittal Plane Motion: A Descriptive and Correlational Study in Healthy Volunteers. Life (Basel). 2023 Feb 7;13(2):461. doi: 10.3390/life13020461. PMID 36836818
- [Background] Zarate-Tejero C, Hidalgo-Garcia C, Lucha-Lopez O, Hernandez-Secorun M, Krauss J, Rodriguez-Rubio P. Association between age, sex and cervical and upper cervical rotation tests. Descriptive and correlational study in healthy volunteers. Ther Adv Chronic Dis. 2023 Apr 29;14:20406223231170158. doi: 10.1177/20406223231170158. eCollection 2023. PMID 37152351
- [Background] Gallego-Izquierdo T, Arroba-Diaz E, Garcia-Ascoz G, Val-Cano MDA, Pecos-Martin D, Cano-de-la-Cuerda R. Psychometric Proprieties of a Mobile Application to Measure the Craniovertebral Angle a Validation and Reliability Study. Int J Environ Res Public Health. 2020 Sep 8;17(18):6521. doi: 10.3390/ijerph17186521. PMID 32911612
- [Background] Takasaki H, Hall T, Oshiro S, Kaneko S, Ikemoto Y, Jull G. Normal kinematics of the upper cervical spine during the Flexion-Rotation Test - In vivo measurements using magnetic resonance imaging. Man Ther. 2011 Apr;16(2):167-71. doi: 10.1016/j.math.2010.10.002. Epub 2010 Nov 4. PMID 21055995
- [Background] Williams MA, McCarthy CJ, Chorti A, Cooke MW, Gates S. A systematic review of reliability and validity studies of methods for measuring active and passive cervical range of motion. J Manipulative Physiol Ther. 2010 Feb;33(2):138-55. doi: 10.1016/j.jmpt.2009.12.009. PMID 20170780
- [Background] Youdas JW, Garrett TR, Suman VJ, Bogard CL, Hallman HO, Carey JR. Normal range of motion of the cervical spine: an initial goniometric study. Phys Ther. 1992 Nov;72(11):770-80. doi: 10.1093/ptj/72.11.770. PMID 1409874
- [Background] Kovacs FM, Bago J, Royuela A, Seco J, Gimenez S, Muriel A, Abraira V, Martin JL, Pena JL, Gestoso M, Mufraggi N, Nunez M, Corcoll J, Gomez-Ochoa I, Ramirez MJ, Calvo E, Castillo MD, Marti D, Fuster S, Fernandez C, Gimeno N, Carballo A, Milan A, Vazquez D, Canellas M, Blanco R, Brieva P, Rueda MT, Alvarez L, Del Real MT, Ayerbe J, Gonzalez L, Ginel L, Ortega M, Bernal M, Bolado G, Vidal A, Ausin A, Ramon D, Mir MA, Tomas M, Zamora J, Cano A. Psychometric characteristics of the Spanish version of instruments to measure neck pain disability. BMC Musculoskelet Disord. 2008 Apr 9;9:42. doi: 10.1186/1471-2474-9-42. PMID 18400084
- [Background] Cleland C, Ferguson S, Ellis G, Hunter RF. Validity of the International Physical Activity Questionnaire (IPAQ) for assessing moderate-to-vigorous physical activity and sedentary behaviour of older adults in the United Kingdom. BMC Med Res Methodol. 2018 Dec 22;18(1):176. doi: 10.1186/s12874-018-0642-3. PMID 30577770
- [Background] Rodriguez-Sanz J, Malo-Urries M, Lucha-Lopez MO, Corral-de-Toro J, Gonzalez-Rueda V, Lopez-de-Celis C, Perez-Bellmunt A, Hidalgo-Garcia C. Is Cervical Stabilization Exercise Immediately Effective in Patients with Chronic Neck Pain and Upper Cervical Spine Dysfunction? Randomized Controlled Trial. Life (Basel). 2022 May 11;12(5):714. doi: 10.3390/life12050714. PMID 35629381
- [Background] Sarig Bahat H, Weiss PL, Sprecher E, Krasovsky A, Laufer Y. Do neck kinematics correlate with pain intensity, neck disability or with fear of motion? Man Ther. 2014 Jun;19(3):252-8. doi: 10.1016/j.math.2013.10.006. Epub 2013 Nov 9. PMID 24291364
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Akodu AK, Akinbo SR, Young QO. Correlation among smartphone addiction, craniovertebral angle, scapular dyskinesis, and selected anthropometric variables in physiotherapy undergraduates. J Taibah Univ Med Sci. 2018 Oct 5;13(6):528-534. doi: 10.1016/j.jtumed.2018.09.001. eCollection 2018 Dec. PMID 31435373